CLINICAL TRIAL: NCT01734863
Title: Post-operative Radiotherapy Randomization in Poor Responders Ewing's Sarcoma Patients
Brief Title: Post-operative Radiotherapy in Poor Responders Ewing's Sarcoma Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHE-BoneT002
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2012-11

CONDITIONS: Ewing's Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy Arm (Experimental): this study arm will take External Beam radiotherapy as follows :
  * Radiotherapy Technique: Conformal radiotherapy, Intensity modulated radiotherapy [IMRT] is allowed.
  * Radiotherapy Dose: 45 Gy/25 fractions/5 weeks (1.8 Gy/fraction). , the inclusion criteria are as following:
    1. Age < 18 years old.
    2. Non-metastatic Ewing Sarcoma patients who will undergo surgery and show poor histologic response to neo-adjuvant chemotherapy.
    3. Negative surgical margins.
    4. Patients show good safety profile and acceptable performance status.
  Interventions: Radiation: External Beam Radiotherapy
- No Radiotherapy Arm (No Intervention): this arm will not take radiotherapy and their inclusion criteria as following:
  1. Age < 18 years old.
  2. Non-metastatic Ewing Sarcoma patients who will undergo surgery and show poor histologic response to neo-adjuvant chemotherapy.
  3. Negative surgical margins.
  4. Patients show good safety profile and acceptable performance status.

INTERVENTIONS:
Radiation: External Beam Radiotherapy
  Arms: Radiotherapy Arm

SUMMARY:
Local recurrence after surgical resection is a complex phenomenon. An important predictive factor is the response to chemotherapy. Central site of disease may be a second independent predictive factor (Lin et al. 2007). Patients with more than 10% viable tumour cells at surgery following neo-adjuvant chemotherapy had a less favourable outcome with an Event-free Survival [EFS] of 47% after 10 years. Patients with good histological response (< 10% viable tumour cells) after chemotherapy alone had a prognosis of about 70% after 10 years.

However, further studies are necessary to determine the merit of adjuvant radiation for high-risk patients (poor responders). Taking into consideration that the toxicity and morbidity of combined surgery and radiation is greater than either alone and must be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old.
* Non-metastatic Ewing Sarcoma patients who will undergo surgery and show poor histologic response to neo-adjuvant chemotherapy.
* Negative surgical margins.
* Patients show good safety profile and acceptable performance status.

Exclusion Criteria:

* Patients who show progressive disease and undergo surgery before the time of local control.
* Patients who undergo Amputation or Rotationplasty will be excluded.
* Post-surgical complications that may hinder the administration of radiotherapy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
improved Local Relapse-free Survival (LRFS) | five year event free survival
  Determine whether the administration of post-operative radiotherapy for poor responder Ewing Sarcoma patients to neo-adjuvant chemotherapy and radical surgery, leads to improved Local Relapse-free Survival (LRFS).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed s zaghloul, MD, Principal Investigator — Children's Cancer Hospital Egypt 57357
Locations (1):
- Children's Cancer Hospital Egypt 57357, Cairo, Egypt